CLINICAL TRIAL: NCT06753682
Title: Effect of the Healthy Plant-based Dietary Pattern As an Adjunct to Non-surgical Periodontal Treatment in Periodontitis: a Randomized Controlled Clinical Trial
Brief Title: Healthy Plant-based Diet and Periodontal Treatment
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Deng Ke Coral, Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UW 24-003
Record Dates: First submitted 2024-12-08; First posted 2024-12-31 (Actual); Last update posted 2024-12-31 (Actual); Status verified 2024-09

CONDITIONS: Periodontal Diseases; Periodontitis; Diet
MeSH Terms: conditions — Periodontal Diseases; Periodontitis

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Healthy Plant Based Diet Group (Experimental): Participants will receive dietary intervention on top of non-surgical periodontal treatment
  Interventions: Behavioral: Healthy Plant Based Diet
- Control Group (No Intervention): Participants will just receive non-surgical periodontal treatment

INTERVENTIONS:
Behavioral: Healthy Plant Based Diet — Registered Dietician will assist in modifying the patient's diet
  Arms: Healthy Plant Based Diet Group

SUMMARY:
Background:

Periodontitis is a highly prevalent chronic disease, affecting around 743 million people globally. In Hong Kong, over 90% of adults have bleeding gums, and 50% of the elderly have severe periodontitis.

The causes of periodontitis are complex, involving polymicrobial dysbiosis, chronic inflammation, immune response, and environmental factors. Current treatments focus on oral hygiene, biofilm/calculus removal, and surgery for advanced cases. While lifestyle and risk factor modifications can improve treatment outcomes, only a few modifiable factors, like smoking cessation and diabetes control, have been established. Identifying more modifiable risk factors and implementing effective interventions are crucial to address this significant public health issue.

Diet has shown to be a major modifiable risk factors in pathophysiology of diabetes mellitus and cardiovascular diseases. The recent Global Burden of Diseases (GBD) study also supports this by pointing out the key dietary risk factors for chronic diseases and mortality. Nonetheless, the role of dietary intervention in the field of periodontitis is poorly understood.

The evidence of a plant-based dietary pattern, defined by a higher consumption of plant foods and lower intake of animal foods, on preventing and treating NCDs is emerging and a "healthy plant-based dietary pattern" is shown to lower risk of periodontitis and elevated serum antibody levels against periodontopathogens. "Healthful plant-based dietary pattern" mainly comprises of high consumption of healthy plant food (e.g., whole grains, fruit and vegetable), but low proportion intake of unhealthy plant food (e.g., refined grains, fruit juices, and sugar-sweetened beverages) .

Although the cross-sectional data from National Health and Nutrition Examination Survey (NHANES) shows promising benefits of the healthful plant-based diet, it is still inconclusive whether "healthful plant-based dietary pattern" is beneficial in preventing and treating periodontal disease. Therefore, it is planned to carry out a high quality, randomised controlled trial to support advocating this dietary pattern in periodontal patients.

Hypothesis:

It is hypothesized that non-surgical periodontal treatment (NSPT) performed in conjunction with healthful plant-based diet would provide additional clinical, immunological and microbiological benefits without incurring malnutrition periodontitis patients

Materials and Methods:

1. Recruitment of subjects

   1. Patients diagnosed with Stage II and Stage III Periodontitis will be recruited from the Reception and Primary Care Clinic of the Prince Philip Dental Hospital and the Institute for Advanced Dentistry, The University of Hong Kong.
   2. Participants enrolled will be randomized into two groups, one test group and one control group (with or without dietary intervention on healthy plant-based diet)
2. Study Procedures

   1. Baseline examination At baseline, besides the routine periodontal examination, patients will undergo dietary assessment by performing the Food Frequency Questionnaire (FFQ), anthropometric measures, oral health related quality of life and physical activity assessment . Biological samples for instance the blood, saliva, fecal and subgingival plaque will also be collected.
   2. Periodontal treatment Step I and Step II periodontal therapy including, oral hygiene instructions, control of risk factors, extraction of hopeless teeth, if any, scaling and root surface debridement will be provided to both groups
   3. Dietary intervention The participants in the test group will participate in a 3-month active intervention phase, a 3-month reinforcement phase, and a 6-month maintenance phase, with the intervention delivered by a trained and registered dietitian. The participants in the control group will continue the ad libitum diets based on their current eating habits and receive no dietary interventions..
   4. Recall Schedule The follow-up visits will be conducted at 2 weeks, 4 weeks, 3, 6 and 12 months after completion of the debridement.

Significance:

This study will provide local data and explore whether healthful plant-based diet as an adjunct to non-surgical periodontal treatment can improve clinical outcome, and provide scientific evidence of its effect on clinical, immunological and microbiological markers of periodontitis.

This can help us understand more on the relationship of healthful plant-based diet and periodontal diseases, which may eventually provide new perspectives for treatment of patients with periodontitis.

ELIGIBILITY:
Inclusion Criteria:

* Chinese ethnicity aged between 18 and 64;
* Generalized Stage II and Stage III periodontitis;
* at least 10 occluding pairs present;
* Good general health;
* Never-smoker or former smoker who had quit smoking successfully for at least 12 months prior to the screening visit;
* Body mass index (BMI) ranging between 18.5 and 28 kg/m2;
* Self-reported inadequacy of hPBD with the main focus on fresh vegetables (<300 g/day) or/and fruit (<200 g/day) with reference to the Dietary Guidelines for Chinese residents (Society, 2022).

Exclusion Criteria:

* Edentulism
* Presence of any systemic disease or taking medication that can alter the manifestation/outcome of periodontal treatment (e.g., uncontrolled diabetes mellitus, hypertension with use of calcium channel blocker, etc.)
* Pregnancy or intention to become pregnant at any point during the study duration
* Need for antibiotic prophylaxis in the context of dental treatment
* Having received non-steroidal anti-inflammatory medication or antibiotics within the previous 3 months
* Having received professional periodontal treatment (other than supragingival cleaning) within the previous 12 months
* History or clinical manifestation of any eating disorder as determined the International Classification of Diseases
* Presence of any dietary restriction (e.g., adherence to a Mediterranean diet), currently taking nutrient supplements or inability to choose his/her diet
* Having obvious weight change (≥5% of current body weight) over the past 6 months
* Participation in another intervention trial
* Inability or unwillingness of individual to give written informed consent

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Changes of Probing pocket depth (PPD) at 6 months after NSPT compared to baseline assessment | 6 months after NSPT

SECONDARY OUTCOMES:
Changes of PPD at 3, 12 months after NSPT compared to baseline assessment | 3 months and 12 months
Changes of Clinical attachment level (CAL) assessed using periodontal probing method at 3, 6 and 12 months after NSPT compared to baseline assessment | 3, 6 and 12 months after NSPT
Changes of the percentage of Bleeding on probing (BOP) assessed using periodontal probing method compared to baseline assessment | 3, 6 and 12 months after NSPT
Changes in subgingival microbiome assessed using 16S rRNA Gene Sequencing at 3, 6 and 12 months after NSPT compared to baseline assessment | 3, 6 and 12 months after NSPT compared to baseline assessment
Changes in gut microbiome assessed using 16S rRNA Gene Sequencing at 3, 6 and 12 months after NSPT compared to baseline assessment | 3, 6 and 12 months after NSPT compared to baseline assessment
Changes in salivary and blood-based biomarker levels at 3, 6 and 12 months after NSPT compared to baseline assessment | 3, 6 and 12 months after NSPT compared to baseline assessment
Changes in healthful plant-based diet index (hPDI) with higher scores indicating a healthier diet at 3,6 and 12 months after NSPT compared to baseline assessment | 3,6 and 12 months after NSPT compared to baseline assessment

CONTACTS AND LOCATIONS:
Locations (1):
- Prince Philip Dental Hospiral, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Li A, Qiu B, Goettsch M, Chen Y, Ge S, Xu S, Tjakkes GE. Association between the quality of plant-based diets and periodontitis in the U.S. general population. J Clin Periodontol. 2023 May;50(5):591-603. doi: 10.1111/jcpe.13785. Epub 2023 Feb 13. PMID 36734066
- [Background] Kassebaum NJ, Bernabe E, Dahiya M, Bhandari B, Murray CJ, Marcenes W. Global burden of severe periodontitis in 1990-2010: a systematic review and meta-regression. J Dent Res. 2014 Nov;93(11):1045-53. doi: 10.1177/0022034514552491. Epub 2014 Sep 26. PMID 25261053
- [Background] Craig WJ, Mangels AR, Fresan U, Marsh K, Miles FL, Saunders AV, Haddad EH, Heskey CE, Johnston P, Larson-Meyer E, Orlich M. The Safe and Effective Use of Plant-Based Diets with Guidelines for Health Professionals. Nutrients. 2021 Nov 19;13(11):4144. doi: 10.3390/nu13114144. PMID 34836399
- [Background] Satija A, Bhupathiraju SN, Rimm EB, Spiegelman D, Chiuve SE, Borgi L, Willett WC, Manson JE, Sun Q, Hu FB. Plant-Based Dietary Patterns and Incidence of Type 2 Diabetes in US Men and Women: Results from Three Prospective Cohort Studies. PLoS Med. 2016 Jun 14;13(6):e1002039. doi: 10.1371/journal.pmed.1002039. eCollection 2016 Jun. PMID 27299701
- [Background] Sanz M, Herrera D, Kebschull M, Chapple I, Jepsen S, Beglundh T, Sculean A, Tonetti MS; EFP Workshop Participants and Methodological Consultants. Treatment of stage I-III periodontitis-The EFP S3 level clinical practice guideline. J Clin Periodontol. 2020 Jul;47 Suppl 22(Suppl 22):4-60. doi: 10.1111/jcpe.13290. PMID 32383274
- [Background] Tonetti MS, Greenwell H, Kornman KS. Staging and grading of periodontitis: Framework and proposal of a new classification and case definition. J Periodontol. 2018 Jun;89 Suppl 1:S159-S172. doi: 10.1002/JPER.18-0006. PMID 29926952
- See also: Related Info — https://www.nature.com/articles/ejcn2011147